CLINICAL TRIAL: NCT01962051
Title: AMPLATZER Cardiac Plug (ACP) Latin American Post Market Observational
Acronym: ACP LA
Status: Withdrawn | Type: Observational
Why Stopped: St. Jude Medical business decision
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL07123
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Delivery system Entry
  Interventions: Device: Amplatzer Cardiac Plug

INTERVENTIONS:
Device: Amplatzer Cardiac Plug

SUMMARY:
The ACP device will be clinically evaluated through a prospective, open-label, nonrandomized, multi-center post market clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented history of paroxysmal, persistent or permanent nonvalvular atrial fibrillation (documentation may include an electrocardiogram (ECG), Holter, or event recorder)
* Subject must have a LAA closure procedure that has already been planned or scheduled by his/her attending physician before entry in the study
* Subject must be greater than or equal to 18 years of age

Exclusion Criteria:

* Subject with an implanted atrial septal defect (ASD) device or patent foramen ovale (PFO) device
* Subject underwent LAA closure procedure prior to study entry (i.e. before signing informed consent
* Subject who has a history of surgical ASD or PFO repair
* Subject with a history of stroke and unrepaired PFO
* Subject who has moderate to severe aortic or mitral valve stenosis or regurgitation requiring surgical or percutaneous intervention as assessed by the Investigator
* Subject who has a mitral or aortic prosthetic valve
* Subject with NYHA grade 4
* Subject with evidence of moderate pericardial effusion at baseline evaluation
* Subject who has complex atheroma with mobile plaque of the descending aorta and/or aortic arch
* Subject who has an intracardiac thrombus
* Subject who has carotid disease as assessed by the Investigator, requiring treatment, which includes revascularization and/or medical treatment
* Subject with active infection or active endocarditis
* Subject who has an acute or recent myocardial infarction (MI) or unstable angina (recent is defined as within 3 months of implant date)
* Subject who has had recent major cardiac surgical procedure (recent is defined as within 6 months of implant date)
* Subject with malignancy or other illness where life expectancy is less than one year
* Subject who is pregnant, breastfeeding, or desires to become pregnant during their first six months of follow-up
* Subject or legally authorized representative who is unable to provide informed consent
* Subject who will not be able to be followed for the duration of the clinical study
* Subject with any medical disorder or severe disability that would interfere with completion or evaluation of clinical study results (for example uncontrolled hypertension, uncontrolled diabetes, blood disorder, renal failure, in situ IVC filter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with nonvalvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of the ACP device in closure of the LAA | 2 years post implant
  Defined as absence of flow or flow of ≤3mm jet into the LAA at procedure and at 6 months, 1 year and 2 years as assessed by Transoesophageal Echocardiography (TOE).
The rate of occurrence for any reported adverse event experienced by subjects enrolled | Through 2 years

IPD SHARING:
Plan to Share IPD: No
No data collected as study stopped before sites activated